CLINICAL TRIAL: NCT02176356
Title: Patient Satisfaction Study of Combined Facial Treatment With BOTOX® Cosmetic, JUVÉDERM® and LATISSE® (HARMONY Study)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: GMA-CMB-14-001
Record Dates: First submitted 2014-06-25; First posted 2014-06-27 (Estimated); Results first posted 2016-06-16 (Estimated); Last update posted 2019-01-09 (Actual); Status verified 2018-12

CONDITIONS: Facial Rhytides; Crow's Feet Lines; Glabellar Lines; Nasolabial Fold
MeSH Terms: interventions — Botulinum Toxins, Type A; Bimatoprost

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- All Participants (Other): JUVÉDERM® ULTRA XC and/or JUVÉDERM® ULTRA PLUS XC and/or JUVÉDERM® VOLUMA® XC injection into facial areas, volume as determined by the investigator on Day 1 with additional treatment at Day 14 if applicable. LATISSE® 1 drop applied to upper eyelid at the base of the eyelashes once daily in the evening for 17 weeks beginning on Day 1. BOTOX® Cosmetic 20U total dose per treatment to glabellar areas and/or 24U total dose per treatment to crow's feet line areas at Month 3.
  Interventions: Biological: onabotulinumtoxinA; Drug: bimatoprost ophthalmic solution 0.03%; Device: JUVÉDERM® ULTRA XC; Device: JUVÉDERM® ULTRA PLUS XC; Device: JUVÉDERM® VOLUMA® XC

INTERVENTIONS:
Biological: onabotulinumtoxinA — onabotulinumtoxinA (BOTOX® Cosmetic) 20U total dose per treatment to glabellar areas and/or 24U total dose per treatment to crow's feet line areas.
  Other Names: botulinum toxin Type A
Drug: bimatoprost ophthalmic solution 0.03% — bimatoprost ophthalmic solution 0.03% (LATISSE®) 1 drop applied to the upper eyelid at the base of eyelashes once daily in the evening for 17 weeks.
  Other Names: LATISSE®
Device: JUVÉDERM® ULTRA XC — JUVÉDERM® ULTRA XC, a hyaluronic acid gel implant (dermal filler), volume injected determined by the investigator.
Device: JUVÉDERM® ULTRA PLUS XC — JUVÉDERM® ULTRA PLUS XC, a hyaluronic acid gel implant (dermal filler), volume injected determined by the investigator.
Device: JUVÉDERM® VOLUMA® XC — JUVÉDERM® VOLUMA® XC, a hyaluronic acid gel implant (dermal filler), volume injected determined by the investigator.

SUMMARY:
A study to evaluate patient satisfaction, aesthetic and psychological impact of combined treatment with BOTOX® Cosmetic (onabotulinumtoxinA), JUVÉDERM® ULTRA XC, JUVÉDERM® ULTRA PLUS XC, JUVÉDERM® VOLUMA® XC, and LATISSE® (bimatoprost ophthalmic solution).

ELIGIBILITY:
Inclusion Criteria:

* Qualified to receive treatment with BOTOX® Cosmetic, a facial filler (JUVÉDERM® ULTRA XC and/or JUVÉDERM® ULTRA Plus XC and/or JUVÉDERM® VOLUMA® XC) and LATISSE® treatment
* Naïve to botulinum toxin therapy of any serotype for any indication
* Naïve to prescription eyelash growth products of any type
* Naïve to dermal filler treatment in the face and neck

Exclusion Criteria:

* Undergone facial plastic surgery, tissue grafting, tissue augmentation or facial dermal filler injections
* Had laser, photomodulation, intense pulsed light, radio frequency, dermabrasion or chemical peel in the face or neck
* Have received skin resurfacing (laser, photomodulation, intense pulsed light, radio frequency, dermabrasion, chemical peel, or non-ablative procedures) in the face or neck within 3 months
* Systemic retinoid therapy within 1 year prior to study enrollment
* Presence of inflammation at the proposed injection site(s)
* Profound atrophy/excessive weakness of muscles in target areas of injection
* Known immunization or hypersensitivity to any botulinum toxin serotype
* Undergone oral surgery or dental procedures within 30 days
* No visible eyelashes
* Use of permanent eyeliner, eyelash implants, semi-permanent eyelash tint, dye or extension
* Use of prescription eyelash growth products
* Unwilling or unable to remove contact lenses prior to study medication application in the evening and keep lenses out for 30 minutes
* Diagnosis of myasthenia gravis, Eaton-Lambert Syndrome, amyotrophic lateral sclerosis, or any other disease that might interfere with neuromuscular function.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2014-06-30 (Actual); Primary Completion 2015-05-03 (Actual); Study Completion 2015-05-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Los Angeles, California, United States

REFERENCES:
- [Background] Weinkle SH, Werschler WP, Teller CF, Sykes JM, Shamban A, Rivkin A, Narurkar VA, Kaminer MS, Dayan S, Cohen JL, Gallagher CJ. Impact of Comprehensive, Minimally Invasive, Multimodal Aesthetic Treatment on Satisfaction With Facial Appearance: The HARMONY Study. Aesthet Surg J. 2018 Apr 6;38(5):540-556. doi: 10.1093/asj/sjx179. PMID 29244069

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Participants
Started | 116
Eligible and Received Treatment | 100
Completed | 93
Not Completed | 23
Not completed — Screen Failure | 14
Not completed — Lost to Follow-up | 4
Not completed — Personal Reasons | 3
Not completed — Other Miscellaneous Reasons | 2

BASELINE CHARACTERISTICS:
Population: Safety population included all enrolled participants who received any study treatment.
Arm/Group | All Participants
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.5 (7.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Satisfaction With Facial Appearance Overall Using a 10-item Questionnaire
Description: Participants assessed their satisfaction with the way they look right now with their entire face in mind using a 10-item questionnaire. Possible responses to each question were: 1=Very dissatisfied, 2=Somewhat dissatisfied, 3-=Somewhat satisfied and 4=Very satisfied. The responses were added across items and transformed to a Rasch scale ranging from 0 (worst) to 100 (best). A positive change from Baseline indicates improvement.
Time Frame: Baseline, Month 4
Population: Modified Intent-to-Treat (mITT) population included all participants who received all 3 treatments and had a Baseline and at least 1 post-treatment efficacy assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 93
score on a scale
  Baseline | 41.22 (11.97)
  Change from Baseline at Month 4 | 31.70 (20.00)

2. Secondary Outcome: Change From Baseline in Aging Appearance Using a 7-item Questionnaire
Description: Participants rated how they look now using a 7-item questionnaire. Possible responses for each question are 1=Definitely disagree, 2=Somewhat disagree, 3=Somewhat agree or 4=Definitely agree. The responses were added across items and transformed to a Rasch score ranging from 0 (worst) to 100 (best). A positive change from Baseline indicates improvement.
Time Frame: Baseline, Month 4
Population: mITT population included all participants who received all 3 treatments and had a Baseline and at least 1 post-treatment efficacy assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 93
score on a scale
  Baseline | 45.07 (18.85)
  Change from Baseline at Month 4 | 28.47 (21.47)

3. Secondary Outcome: Change From Baseline in Age Appraisal Using a Visual Analogue Scale (VAS)
Description: Participants assessed how old they think they look compared to their actual age using a VAS by placing a mark on a number on a horizontal line where the far left of the line= -15 (look 15 years younger), 0=look current age, to the far right of the line=15 (look 15 years older). A positive change from Baseline indicates improvement.
Time Frame: Baseline, Month 4
Population: Participants from the mITT population, all participants who received all 3 treatments and had a Baseline and at least 1 post-treatment efficacy assessment, with data available for analysis.
Measure: Mean (Standard Deviation); unit: years
Arm/Group | All Participants
Number analyzed (Participants) | 93
years
  Baseline | 0.1 (4.28)
  Change from Baseline at Month 4 (n=92) | -4.6 (4.36)

4. Secondary Outcome: Change From Baseline in Social Confidence Using an 8-item Questionnaire
Description: Participants assessed their social confidence with their facial appearance in mind in the past week using an 8-item questionnaire. Possible responses for each question are 1=Definitely disagree, 2=Somewhat disagree, 3=Somewhat agree or 4= Definitely agree. The responses were added across items and transformed to a Rasch score ranging from 0 (worst) to 100 (best). A positive change from Baseline indicates improvement.
Time Frame: Baseline, Month 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 93
score on a scale
  Baseline | 62.70 (21.74)
  Change from Baseline at Month 4 | 18.24 (23.04)

5. Secondary Outcome: Change From Baseline in Psychological Well-Being Using a 10-item Questionnaire
Description: Participants assessed their psychological well-being with their facial appearance in mind using a 10-item questionnaire. Possible responses for each question are 1=Definitely disagree, 2=Somewhat disagree, 3=Somewhat agree or 4= Definitely agree. The responses were added across items and transformed to a Rasch score ranging from 0 (worst) to 100 (best). A positive change from Baseline indicates improvement.
Time Frame: Baseline, Month 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 93
score on a scale
  Baseline | 62.78 (22.45)
  Change from Baseline at Month 4 | 19.89 (20.63)

6. Secondary Outcome: Participant's Self- Perception of Age (SPA)
Description: Participants assessed SPA by answering the question: How do you think your facial appearance looks compared to your age today? Participants recorded how many years younger or older they thought their facial appearance made them look. A negative result indicates improvement (a younger appearance).
Time Frame: Baseline, Month 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: years
Arm/Group | All Participants
Number analyzed (Participants) | 93
years
  Baseline | 0.2 (4.08)
  Month 4 | -4.6 (4.19)

7. Secondary Outcome: Change From Baseline in Investigator's Assessment of Severity of Glabellar Lines (GLs) at Maximum Frown Using the Facial Wrinkle Scale (FWS)
Description: The investigator assessed the severity of the participant's GLs using the 4-point FWS where: 0=None, 1=Mild, 2=Moderate or 3=Severe. A negative change from Baseline indicates improvement.
Time Frame: Baseline, Month 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 89
score on a scale
  Baseline | 2.6 (0.50)
  Change from Baseline at Month 4 | -1.6 (0.78)

8. Secondary Outcome: Change From Baseline in Investigator's Assessment of the Severity of Crow's Feet Lines (CFLs) at Maximum Smile Using the FWS
Description: The investigator assessed the severity of the participant's CFLs using the 4-point FWS where: 0=None, 1=Mild, 2=Moderate or 3=Severe. A negative change from Baseline indicates improvement.
Time Frame: Baseline, Month 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 90
score on a scale
  Left_Baseline | 2.5 (0.50)
  Left_Change from Baseline at Month 4 | -1.0 (0.85)
  Right_Baseline | 2.5 (0.50)
  Right_Change from Baseline at Month 4 | -1.0 (0.85)

9. Secondary Outcome: Change From Baseline in Investigator's Global Eyelash Assessment Score (GEAS)
Description: The investigator assessed the participant's eyelash prominence using the 4-point GEAS where: 1=Minimal (worst), 2=Moderate, 3=Marked and 4=Very Marked (best). A positive change from Baseline indicates improvement.
Time Frame: Baseline, Month 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 93
score on a scale
  Baseline | 1.8 (0.42)
  Change from Baseline at Month 4 | 1.5 (0.65)

10. Secondary Outcome: Change From Baseline in the Investigator's Assessment of the Participant's Overall Mid-Face Volume Deficit Using the 6-Point MFVDS
Description: The investigator assessed overall mid-face volume deficit using the Mid-face Volume Deficit Scale (MFVDS) where: 0=None (moon face; fullness) [best], 1=Minimal (flattening), 2=Mild (mild concavity), 3=Moderate (moderate concavity, 4=Significant (significant concavity) and 5=Severe (wasting) [worst]. A negative change from Baseline indicates improvement.
Time Frame: Baseline, Month 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 89
score on a scale
  Baseline | 3.1 (0.36)
  Change from Baseline at Month 4 | -1.7 (0.80)

11. Secondary Outcome: Change From Baseline in the Investigator's Assessment of the Participant's Nasolabial Folds Severity
Description: The investigator assessed the participants nasolabial folds severity using the 5-Point Nasolabial Fold Severity (NLFS) Scale where: 0=None (no wrinkles) [best], 1=Mild (shallow, just perceptible wrinkle), 2=Moderate (moderately deep wrinkle), 3=Severe (deep wrinkle) or 4= Extreme (very deep wrinkle). A negative change from Baseline indicates improvement.
Time Frame: Baseline, Month 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 90
score on a scale
  Baseline | 2.6 (0.51)
  Change from Baseline at Month 4 | -1.0 (0.85)

12. Secondary Outcome: Change From Baseline in the Investigator's Assessment of the Participant's Oral Commissures Severity
Description: The investigator assessed the participant's oral commissure using the 4-Point Oral Commissure Severity Scale (OCSS) where: 0=None, 1=Mild, 2=Moderate or 3=Severe. A negative change from Baseline indicates improvement.
Time Frame: Baseline, Month 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 86
score on a scale
  Baseline | 2.1 (0.49)
  Change from Baseline at Month 4 | -0.9 (0.67)

13. Secondary Outcome: Change From Baseline in the Investigator's Assessment of the Participant's Perioral Lines Severity
Description: The investigator assessed the participant's perioral lines severity using the 4-Point Perioral Lines at Rest Severity Scale (POLSS) where: 0=None (no lines) [best], 1=Mild (few, shallow lines), 2=Moderate (some moderate lines) or 3=Severe (many deep lines or crevices)[worst]. A negative change from Baseline indicates improvement.
Time Frame: Baseline, Month 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 59
score on a scale
  Baseline | 2.0 (0.57)
  Change from Baseline at Month 4 | -1.1 (0.68)

14. Secondary Outcome: Change From Baseline in the Participant Satisfaction With Appearance of Periorbital Area
Description: Participants assessed how their overall eye appearance has affected them over the past 7 days using the 9-item Periorbital Aesthetic Appearance Questionnaire (PAAQ). Possible responses to each question were: 0=Never (best), 1=Rarely, 2=Some of the time, 3=Most of the time and 4=All of the time with a total possible score of 0 to 36. A negative change from Baseline indicates improvement.
Time Frame: Baseline, Month 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 93
score on a scale
  Baseline | 21.1 (6.71)
  Change from Baseline at Month 4 | -12.6 (7.61)

ADVERSE EVENTS:
Description: The Safety population, all enrolled participants who received treatment with any study drug, was used to determine the number of participants at risk for Serious Adverse Events and Non-Serious Adverse Events.
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/100
Other Adverse Events (participants affected / at risk) | 18/100
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=100)
Contusion (Injury, poisoning and procedural complications) | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.